CLINICAL TRIAL: NCT05804695
Title: Arthroscopic Temporomandibular Joint Disc Repositioning
Brief Title: Evaluation of the Arthroscopic Temporomandibular Joint Disc Repositioning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Future University in Egypt (Other)
Responsible Party: Principal Investigator, Medhat Sameh Abdelaziz, Assistant Lecturer of Prosthodontics, Future University in Egypt
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FUE.REC (9)/1-2020
Record Dates: First submitted 2023-03-27; First posted 2023-04-07 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-03

CONDITIONS: Temporomandibular Joint Disc Displacement

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arthroscopic Temporo-mandibular joint disc repositioning under General anathesia (Experimental)
  Interventions: Procedure: Arthroscopic TMJ disc repositioning under GA

INTERVENTIONS:
Procedure: Arthroscopic TMJ disc repositioning under GA — a surgical procedure used to treat Tempro- mandibular disc displacement using arthroscope.

SUMMARY:
1. Full medical and dental history will be taken from the patient participating in this study.
2. A written consent to be signed by the patient for the potentials of operative and postoperative complications.
3. The skin is prepared by antiseptic solution then surgical drapes exposing the ear lobule and the outer canthus of the eye. The entry point at maximum convexity of glenoid fossa with palpation technique for primary arthroscopy technique , diagnostic sweep followed by second puncture using triangulation technique
4. Discopexy technique to be performed with the following steps : anterior release , disc reduction, retro-discal scarification, and disc fixation using ligature wire and button.
5. The trocar then observed on the monitor entering the joint space. Once intra-articular, the trocar should be removed, and drainage of the irrigating fluid through the cannula.
6. A hook probe is inserted through the operative cannula. The intra-articular incision begins at the juncture between the pterygoid shadow and the anterior recess then myotomy to the lateral pterygoid muscle is done.
7. The operative cannula then "walked back" in the lateral sulcus to the posterior pouch. The condyle should be pulled forward. The disc then reduced by compressing the retrodiscal tissue laterally and inferiorly with a straight probe, with the condyle in a forward or forward and contralateral position.
8. Next, Disc fixation should be accomplished using ligation wire. The target area of fixation is the posterior lateral corner of the disc. A suitable gauge needle with a single wire inserted through the skin and subcuticular tissues, touching the condylar head, into the inferior joint space, and then angled superiorly. Once that completed, a straight Meniscus Mender II inserted in the preauricular skin crease 5 to 7 mm below the fossa portal into the superior joint space.
9. The snare of the Meniscus Mender was then inserted through the Meniscus Mender cannula, and the ligation wire then passed through the 20-gauge needle anteriorly and caught by the snare to have both ends of the suture exited the skin.
10. Small skin incisions should be done at the exit points of the wire superiorly with a no. 11 blade through the skin and subcutaneous tissue. A straight hemostat used to dissect down, tracing anteriorly to the capsule along the course of the facial nerve. Posteriorly, the dissection continued down halfway to the capsule.
11. A suitable gauge needle then used to pass the anterior wire through the slit incision, deep to the capsule, and back out to the posterior slit incision, so that both free ends of the ligation wire exiting posteriorly through the posterior slit incision. With the disc held in reduction, a tight surgeon's knot tied plicating the disc to the lateral capsule and holding the disc in a posterior lateral position and buttons then used.
12. Finally, the arthroscope used to check the position of the disc under function9.
13. Postoperative instructions and medications :

    * Analgesics
    * Antibiotic coverage
    * MRI 6 months postoperative to assess disc reduction
    * Follow up appointment one week, one month ,three months and 6 months (Buttons will be removed two weeks postoperatively) To assess the disc position and testing for any facial nerve affection Then, measurements of the maximum mouth opening in millimeters.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of TMJ disorder (Pain, limitation and/or locking)
* Unilateral or bilateral TMJ internal derangement Wilkes stage III, IV
* Failed Conservative treatment for two months if it was indicated
* Age between 20- 50 years old

Exclusion Criteria:

* Systemic Disease such as uncontrolled Diabetes, uncontrolled hypertension
* Patient who had a previous Intracapsular TMJ surgery
* Tumors and TMJ ankylosis
* Edentulous patients

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2020-02-20 (Actual); Primary Completion 2023-03-20 (Actual); Study Completion 2023-03-25 (Actual)

PRIMARY OUTCOMES:
Change in the measurements of the maximum inter-incisal opening (MIO) | pre surgery and after 6 months from surgery
  Change in the measurements of the maximum inter-incisal opening (MIO) in millimeter measured by a ruler preoperatively and postoperatively in the follow up appointments.

CONTACTS AND LOCATIONS:
Locations (1):
- Future University in Egypt, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided